CLINICAL TRIAL: NCT01029496
Title: Effect of Umbilical Cord Clamping Time on Newborns
Brief Title: Immediate VS Delayed Cord Clamping on Newborns
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hainan Medical College (Other)
Responsible Party: huangyuanhua, hainan medical college
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: hainanmc
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2009-09

CONDITIONS: Newborn; Umbilical Cord
Keywords: umbilical CORD CLAMPING; Neonatal anemia; Omphalitis
MeSH Terms: conditions — Anemia, Neonatal | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: different time of umbilical cord clamping — 1. for normal birth(apgar score over 7),include:term ,preterm,normal birth or cesarean section : experimental group1: waiting until the ceased of the umbilical cord pulsing, then cut the cord.before cutting the cord, the baby is keeping warm and put over mother's abdomen.
     control group 1-1: clamping and cut the cord within 10 second after birth. control group1-2: clamping and cut the cord 90 second after birth.
  2. for in case of asphyxia(regardless term or preterm,normal birth or cesarean section born):
  experimental group2: resuscitate on bed site with the cord unclamped until the umbilical cord ceased pulsing.
  control group 2-1 clamping and cut the cord within 10 second. and resuscitate the baby after transfer to the Irradiation table.
  Other Names: DELAYED CORD CLAMPING AND IMMIDIATE CORD CLAMPING

SUMMARY:
The best time of the umbilical cord clamping has not been fully understood. immediate cord clamping (with in 10 seconds after birth) has been standardized practice for many years, while WHO protocol recommends to wait for 60-90 seconds. but the umbilical cord may still pulse for more than 90 seconds. is it best to wait longer until the pulsing ceased? how the time of umbilical cord will affect the newborn? will the longer time be less umbilical bleeding and shorter departure time of the cord? the hypothesis of this study is: to cut the cord after the pulsing ceased is the best time for cord clamping and will result in better quality of life for the newborn and less cord bleeding and earlier departure time of the cord, that means less infections of the cord.

DETAILED DESCRIPTION:
1. for normal newborn (apgar score over 7), regardless term or preterm,normal birth or cesarean section born: experimental group1: waiting for the ceased of the umbilical cord pulsing, then cut the cord.before cutting the cord, the baby is keeping warm and put over mother's abdomen.

   control group 1-1: clamping and cut the cord within 10 second after birth. control group1-2: clamping and cut the cord 90 second after birth.
2. for in case of newborn asphyxia(regardless term or preterm,normal birth or cesarean section born):

experimental group2: resuscitate on bed site with the cord unclamped until the umbilical cord ceased pulsing.

control group 2-1 clamping and cut the cord within 10 second. and resuscitate the baby after transfer to the Irradiation table.

ELIGIBILITY:
Inclusion Criteria:

* all living baby after birth, including term, preterm, normal birth, cesarean section, apgar score over 7 or less than that.

Exclusion Criteria:

* still birth

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
hemoglobin level of the baby 1 month after birth | 2 years

SECONDARY OUTCOMES:
departure time of the umbilical cord | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: hua shao ping, professor, Study Director — director of ob&gny dpt.of appendix hospital of hainan medical college
Locations (1):
- Hainan Medical College Appendix Hospital, Haikou, Hainan, China

REFERENCES:
- [Background] zhang hong-yu,Meng li-ping,Xie chun-li.summary of current clinical protocols of umbilical cord care.Chinese journal of nurisng.3(43):275-277,2008